CLINICAL TRIAL: NCT00002740
Title: Phase I Pilot Study of Multiple Cycles of High Dose Chemotherapy With Peripheral Blood Stem Cell Infusions In Advanced Stage Neuroblastoma
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation Followed by Surgery and/or Radiation Therapy in Treating Young Patients With Advanced Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 3951; CCG-3951 (Other: Children's Cancer Group); CDR0000064656 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Platinum; Cyclophosphamide; Doxorubicin; Etoposide; Mesna; Vincristine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment - Carboplatin Chemotherapy (Experimental): See detailed description.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: mesna; Drug: vincristine sulfate; Procedure: conventional surgery; Procedure: peripheral blood stem cell transplantation; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Biological: filgrastim
  Other Names: G-CSF (Granulocyte colony stimulating factor; Neupogen; NSC# 614629
Drug: carboplatin
  Other Names: CBDCA; Cis-diamine [1,1-cyclobutane-dicarboxylato] platinum); NSC# 241240
Drug: cyclophosphamide
  Other Names: Cytoxan; CTX; NSC# 26271
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin; NSC #123127
Drug: etoposide
  Other Names: VP-16; NSC# 141540
Drug: mesna
  Other Names: Sodium 2-mercaptoethane sulfonate; NSC# 113891
Drug: vincristine sulfate
  Other Names: Oncovin; VCR; Leucocristine; NSC# 67474
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy drugs and kill more tumor cells. Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy plus peripheral stem cell transplantation followed by surgery and/or radiation therapy in treating young patients who have newly diagnosed advanced neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the maximum tolerated dose of carboplatin that can be given in combination with cyclophosphamide (CTX) and etoposide following high dose CTX, doxorubicin, and vincristine in patients with newly diagnosed stage IV neuroblastoma. II. Determine the hematologic and nonhematologic toxic effects of this regimen in this patient population. III. Determine the change in neuroblastoma tumor cell content in peripheral blood stem cells (PBSC) collected following chemotherapy. IV. Assess the feasibility of repetitive collection, storage, and infusion of PBSC with multicycle high-dose chemotherapy in pediatric patients. V. Assess hematopoietic recovery following PBSC infusion as well as the CD34 content and CFU-GM yield of the PBSC products. VI. Assess the response rate and disease-free survival in the context of a phase I pilot study. VII. Determine the feasibility of administering twice-daily radiotherapy fractions to post-chemotherapy residual tumor volumes in neuroblastoma patients.

OUTLINE: This is a dose escalation study of carboplatin. Patients receive induction chemotherapy consisting of vincristine IV over 24 hours, cyclophosphamide IV over 4 hours, and doxorubicin IV over 24 hours on days 0, 1, 21, and 22. Patients receive filgrastim (G-CSF) subcutaneously (SQ) or IV beginning on days 3 and 24 and continuing until blood counts recover. Patients undergo peripheral blood stem cell (PBSC) collection after course 2 of induction chemotherapy. Patients receive G-CSF SQ or IV for 2 days prior to and during collection. PBSC are collected daily for 1-3 days. Patients may undergo autologous bone marrow collection after course 1 of consolidation therapy (after PBSC collection). Following mobilization, patients receive consolidation chemotherapy consisting of etoposide IV over 4 hours on days 0, 1, and 2 and carboplatin IV over 1 hour and cyclophosphamide IV over 4 hours on days 0 and 1. Patients receive G-CSF SQ or IV beginning on day 3 (within 4 hours of PBSC infusion) and continuing until blood counts recover. Patients receive PBSC reinfusion at 48-72 hours following completion of each chemotherapy course. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Upon recovery from consolidation chemotherapy, patients with no disease progression undergo tumor resection with or without radiotherapy. Patients undergoing radiotherapy receive therapy twice daily over 7 days. Patients with no disease progression, less than 2% detectable bone marrow disease, and adequate bone marrow cellularity may undergo additional therapy consisting of autologous bone marrow transplantation per appropriate transplant protocol. Cohorts of 6-12 patients receive escalating doses of carboplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 or 4 of 12 patients experience dose limiting toxicity. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 24-30 patients will be accrued for this study within approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed stage IV neuroblastoma by one of the following: Histologic verification Demonstration of tumor cell clumps in bone marrow with elevated urinary catecholamine metabolites Initial presentation with low-stage disease allowed if followed by progression to stage IV disease

PATIENT CHARACTERISTICS: Age: 1 to 21 Performance status: Not specified Hematopoietic: (unless bone marrow involvement by tumor) Absolute neutrophil count greater than 1,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 3.0 mg/dL Renal: Creatinine less than 1.5 mg/dL Creatinine clearance or radionuclide GFR greater than 60 mL/min Cardiovascular: EKG normal Ejection fraction at least 55% by radionuclide MUGA OR Fractional shortening at least 28% by echocardiogram Other: No other significant organ dysfunction that precludes study treatment Body weight at least 10 kg Not pregnant or nursing Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: No prior systemic chemotherapy No prior radiotherapy except as emergency treatment

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 1996-05; Primary Completion 2004-03 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Event Free Survival
  Determine the maximum tolerated dose of a combination of cyclophosphamide, carboplatin, and etoposide for 3 consecutive courses following 2 cycles of a fixed dose of high dose cyclophosphamide, doxorubicin, and vincristine given on a 21 day schedule using G-CSF in combination with peripheral blood stem cells.

CONTACTS AND LOCATIONS:
Overall Officials: Susan G. Kreissman, MD, Study Chair — Duke Cancer Institute
Locations (7):
- United States (7):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Bensimhon P, Villablanca JG, Sender LS, Matthay KK, Park JR, Seeger R, London WB, Yap JS, Kreissman SG. Peripheral blood stem cell support for multiple cycles of dose intensive induction therapy is feasible with little risk of tumor contamination in advanced stage neuroblastoma: a report from the Childrens Oncology Group. Pediatr Blood Cancer. 2010 Apr;54(4):596-602. doi: 10.1002/pbc.22344. PMID 20049927